CLINICAL TRIAL: NCT06946758
Title: The Effects of Aerobic Exercise Combined With Core Stabilisation Training on Functional Capacity, Physical Performance and Fall Risk in Geriatric Individuals With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758?
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: chronic low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups; Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group will receive core stabilisation exercises 3 days a week for 8 weeks. Core exercise programme was applied to the patients three days a week for 8 weeks. The programme consisted of two weekly parts, and each part was planned according to the weeks by ordering from easy to difficult. Prior to the core stabilisation exercise programme, low intensity 5-10 min warm-up 30 min core exercises consisting of 3 levels were performed. Exercises progressed from easy to difficult according to the condition of the patients.
  Interventions: Other: Core stabilization exercises
- Aerobic Exercise Group (Experimental): Core stabilisation exercises applied to the control group were applied to the aerobic exercise group. After the core stabilisation exercises, aerobic exercise was performed with a stationary bicycle at a speed of 50 rpm for approximately 40 minutes.
  Interventions: Other: Aerobic Exercises

INTERVENTIONS:
Other: Core stabilization exercises — Patients in the core stabilisation exercise group underwent a total of 24 sessions of core stabilisation exercise programme 3 days a week (with at least 1 day of rest between each session) for a total of 8 weeks. Each exercise session was performed under the supervision of a physician in the Department of Physical Medicine and Rehabilitation, Istanbul University, Istanbul Faculty of Medicine. Each session was arranged as 35-minute programmes with an average of 8-10 patients, 5 minutes of which was warm-up. Before starting the exercise, patients were taught to reduce lumbar lordosis by contracting and drawing in the abdominal muscles and to find a lumbar and pelvic neutral position by moving the pelvis forwards and backwards. In each session, the neutral position was found first and attention was paid to maintain the neutral position throughout the exercise. The exercises consisted of 3 levels. The exercise level was completed gradually
  Other Names: Control Group
  Arms: Control Group
Other: Aerobic Exercises — The aerobic exercise group underwent core stabilisation exercises applied to the control group. After the core stabilisation exercises, aerobic exercise was performed with a stationary bicycle at a speed of 50 rpm for approximately 40 minutes.
  Arms: Aerobic Exercise Group

SUMMARY:
The aim of the study is to evaluate the effects of aerobic exercise combined with core stabilisation training (CSE) in elderly individuals with chronic non-specific low back pain (CNSBP). The effects on functional capacity, quality of life, fall risk, functional status and physical performance will be investigated. Core stabilisation exercises will be applied to both groups. The aerobic exercise intervention group will receive aerobic exercise in addition to core stabilisation exercises. The evaluations will be performed before and after the treatment and the treatment is planned for 3 days a week for 8 weeks. The 6-minute walk test (6MWT) will be used to assess functional capacity, Visual Analogue Scale will be used to assess pain intensity, Oswestry Scale will be used to assess functional status in terms of low back pain, Biodex balance device will be used to assess fall risk, Beck Depression Scale will be used to assess depression, Tampa Kinesiophobia Scale will be used to assess kinesiophobia.

DETAILED DESCRIPTION:
Ageing is associated with a decrease in physiological and functional capacities and quality of life. Guidelines recommend at least 150 minutes of moderate-intensity aerobic activity or 75 minutes of vigorous aerobic activity per week and muscle-strengthening activities at least two days per week. With increasing life expectancy, the risk of major health problems affecting the health and well-being of older adults, such as cardiovascular disease and non-communicable diseases related to inactivity, such as diabetes, cognitive decline and poor mental health, is increasing. Considering the problems accompanying low back pain in elderly individuals, regular aerobic exercise at a moderate pace will have a positive effect on quality of life. Aerobic exercises such as walking and swimming can maintain and improve cardiovascular fitness while providing an effective treatment for various chronic and acute diseases ranging from cardiovascular disease to thrombo-embolic stroke, hypertension, type 2 diabetes mellitus, osteoporosis, obesity, colon cancer, breast cancer, anxiety and depression . Regular light-paced aerobic exercise is a well-established protective factor for the prevention and treatment of non-communicable diseases such as cardiovascular disease, stroke, diabetes, as well as some types of cancer such as breast and colon cancer. In the literature, it has been reported that static stabilisation exercises, dynamic exercises, a general exercise programme including a combination of muscle strength, flexibility and aerobic fitness, progressive aerobic exercise and progressive resistance exercise are effective in chronic nonspecific low back pain and that static stabilisation exercises and dynamic exercises are effective on functional status in addition to pain. Although it is generally reported that aerobic exercise is effective in patients with NSBA, there is no clear information in the literature about which exercise methods are more effective in the treatment of NSBA. In addition, many factors such as compliance of the patient population, education, and social status may affect the type of exercise that can be applied. Therefore, it is important to compare the recommended exercise protocols with various exercise programmes.

In this context, the aim of investigators study was to evaluate the effects of aerobic exercises combined with core exercises on functional status and physical performance in geriatric individuals with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complaints of low back pain for more than 3 months
* Patients aged between 65-84 years
* Patients with a mini-mental status test score above 24

Exclusion Criteria:

* Those with radicular leg pain, sensory and motor deficits in the lower extremities and low back pain with inflammatory character
* Those with previous spinal surgery, spondylolysis, spondylolisthesis, spinal stenosis, vertebral compression, fracture, previous or ongoing spinal infection in past history and examinations

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 8 week
  Visual Analogue Scale (VAS) was used to determine the presence and severity of low back pain in the study participants. GAS is a practical test with high validity and reliability in pain assessment. GAS is an assessment method numbered from 0 to 10, where '0' indicates no pain and '10' indicates the presence of the most severe pain. Participants were asked to mark the degree of pain they had on this scale and recorded.
Disability | 8 week
  Functional status was assessed using the Oswestry Disability Index (ODI). The OSI is a widely used questionnaire for the assessment of functional status in patients with low back pain. It includes subjective assessment. There are items including activities of daily living such as pain intensity, self-care, lifting, walking, sitting, standing, sleeping, social life and travelling information. The items are scored between 0-5. The final score is calculated by taking the patient's score as a percentage of the maximum score. Higher scores indicate an increasing level of disability. Turkish validity and reliability was performed by Yakut et al. in 1998.
Risk of fall | 8 week
  Biodex balance system (Biodex Medical System Inc., NY, USA, Model SW45-30D-E6N, SD 950-304) was used for fall risk assessment. This device creates stability indices by evaluating movements in the overall, anterior-posterior and right-left (medial-lateral) directions. Its validity and reliability have been established in this field. It has static and dynamic modes and 12 mobility levels of the platform (mobility level of the floor). In the limit of stability test, there are 9 balls, 1 in the middle and 8 on the edges, and when these balls light up, the person should move the centre of gravity to the burning ball and keep it there for 0.25 seconds. Each ball flashes once during the test and after the ball on the edge lights up, the ball in the centre lights up again. The aim is to move the centre of gravity in the specified direction. The test was performed three times and the extinguishing time of all balls was recorded by the device.

SECONDARY OUTCOMES:
Cardiopulmonary capacity | 8 week
  The 6-minute walk test is used as a simple measure of aerobic exercise capacity. During this test, you walk at a normal pace for six minutes on a 30-metre long hard surface track, marking the track every 3 metres and placing a cone at the end of the 30-metre track and walking back around it. This test can be used to monitor your response to treatments for heart, lung and other health problems.
Depression | 8 week
  Beck depression scale is a widely used psychological measurement tool to assess depression symptoms. This scale developed by Aaron T. Beck is an important tool used to determine the level of depression of individuals and in treatment processes. Beck depression scale consists of a series of questions including various emotional, cognitive and physical symptoms and the answers to the questions provide information about the severity of depression.
Kinesiophobia | 8 week
  The level of kinesiophobia was evaluated with the 'Tampa Kinesiophobia Scale (TKS)'. The TQS is a 17-question questionnaire developed for musculoskeletal pain, which has been validated and reliable in Turkish. In the scale, a 4-point Likert scoring system (1=Strongly disagree, 2=Agree, 3=Disagree, 4=Strongly agree) is used for each question. As a result of the questionnaire, the person receives a total score between 17-68 according to the answers given. A high score indicates a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, PhD., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Consider briefly explaining why IPD will not or might not be shared.

REFERENCES:
- [Derived] Kuzu S, Canli M, Valamur I, Ozudogru A, Alkan H, Hartavi A. Effects of aerobic exercise in addition to core stabilization exercises on functional capacity, physical performance and fall risk in geriatric individuals with chronic non-specific low back pain. BMC Sports Sci Med Rehabil. 2025 Jul 29;17(1):218. doi: 10.1186/s13102-025-01271-7. PMID 40734175